CLINICAL TRIAL: NCT05133297
Title: A Phase 2A, Randomized, Double-blind, Double-dummy, Tofacitinib-parallel-group Study to Evaluate the Safety and Efficacy of TLL-018 in Active Rheumatoid Arthritis Who Had an Inadequate Response or Intolerance to Methotrexate.
Brief Title: The Safety and Efficacy of TLL-018 in Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Highlightll Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TLL-018-201
Record Dates: First submitted 2021-11-15; First posted 2021-11-24 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): TLL018 tablets, 1piece,BID
  Interventions: Drug: TLL-018
- Sequence 2 (Experimental): TLL018 tablets, 2pieces, BID
  Interventions: Drug: TLL-018
- Sequence 3 (Experimental): TLL018 tablets, 3pieces, BID
  Interventions: Drug: TLL-018
- Sequence 4 (Active Comparator): TOFA tablets, 1pieces, BID
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: TLL-018 — Oral tablets administered at dose1 BID daily for 24 weeks.
  Other Names: Sequence 1
  Arms: Sequence 1
Drug: TLL-018 — Oral tablets administered at dose2 BID daily for 24 weeks.
  Other Names: Sequence 2
  Arms: Sequence 2
Drug: TLL-018 — Oral tablets administered at dose3 BID daily for 24 weeks.
  Other Names: Sequence 3
  Arms: Sequence 3
Drug: Tofacitinib — Oral tablets administered at 5 mg BID daily for 24 weeks.
  Other Names: Sequence 4
  Arms: Sequence 4

SUMMARY:
This is a randomized, double-blind, double-dummy, tofacitinib-parallel-group, phase 2A study to assess the safety and efficacy of TLL-018 in active rheumatoid arthritis subject who had an inadequate response or intolerance to methotrexate.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with RA based on either the 1987-revised American College of Rheumatology (ACR) classification criteria or the 2010 ACR/European League against Rheumatism (EULAR) criteria and have an inadequate response or intolerance to methotrexate.
2. Subjects must have been receiving oral or parenteral methotrexate therapy ≥ 3 months and on a stable prescription of 7.5 to 25 mg/week for at least 4 weeks prior to Baseline Visit.
3. Have active RA as defined by the following minimum disease activity criteria:

   * ≥ 6 swollen joints (based on 66 joint counts) at Screening and Baseline Visits;
   * ≥ 6 tender joints (based on 68 joint counts) at Screening and Baseline Visits;
   * high-sensitivity C-reactive protein (hsCRP) > upper limit of normal (ULN) OR positive for both rheumatoid factor and anti-cyclic citrullinated peptide (CCP) at Screening.
4. For subjects with inadequate response to methotrexate, subjects must have discontinued all oral disease-modifying anti-rheumatic drugs (DMARDs) prior to Baseline Visit as specified below or for at least five times the mean terminal elimination half-life of a drug, whichever is longer:

   * ≥4 weeks prior to Baseline Visit for minocycline, penicillamine, sulfasalazine, hydroxychloroquine, chloroquine, azathioprine, gold formulations, cyclophosphamide;
   * ≥12 weeks prior to Baseline Visit for leflunomide if no elimination procedure was followed, or adhere to a washout procedure (i.e., 11 days washout with colestyramine, or 30 days washout with activated charcoal).
5. The organ function level must meet the following requirements:

Bone marrow: Blood routine results showed hemoglobin ≥90g/L, platelet ≥100×109/L, neutrophil absolute count ≥1.5×109/L; Liver: serum bilirubin ≤1.5 times the upper limit of normal value, aspartate aminotransferase (AST) ≤1.5 times the upper limit of normal value, alanine aminotransferase (ALT) ≤1.5 times the upper limit of normal value; Serum creatinine <1.5 times the upper limit of normal value; Urine protein ≤1+, if urine protein >1+, urine protein should be collected for 24 hours, the total amount should be ≤1 g. Female subjects of childbearing potential must test negative for pregnancy.

Exclusion Criteria:

1. History of Felty syndrome (Rheumatoid arthritis - Splenomegaly syndrome).
2. A history of herpes zoster or disseminated herpes simplex.
3. Treatment with any JAK inhibitor (tofacitinib, baricitinib, ruxolitinib) within 2 weeks prior to study start.
4. Subjects have severe, progressive or uncontrollable symptoms of kidney, liver, blood, gastrointestinal, lung, cardiovascular, neurological or brain disease.
5. Current treatment or treatment within 4 weeks or 5 half-lives (whichever is longer) prior to the first dose of study medication with another investigational medication or current enrollment in another investigational drug protocol.
6. If the laboratory T-Spot test (or other TB diagnostic test) is positive, the investigator will determine the activity based on the history and clinical manifestations, and the patients diagnosed as active TB should be excluded.
7. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody.
8. Pregnant or breastfeeding female.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants American College of Rheumatology 50% (ACR50) Response at Week 12 | Week 12
  A participant was a responder if the following 3 criteria for improvement from baseline were met:
  * ≥50% improvement in 68-tender joint count;
  * ≥50% improvement in 66-swollen joint count; and
  * ≥50% improvement in at least 3 of the 5 following parameters:

SECONDARY OUTCOMES:
Number of Participants American College of Rheumatology 20% (ACR20) Response | Week 4, 8, 12, 16, 20 and 24
  ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in painful and tender joint count; >= 20% improvement in swollen joint count; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP)at each visit.
Number of Participants Achieving American College of Rheumatology 50% (ACR50) Response | Weeks 4, 8, 12, 16, 20 and 24
  ACR50 response: greater than or equal to (>=) 50 percent (%) improvement in painful and tender joint count; >= 50% improvement in swollen joint count; and >= 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP) at each visit.
Number of Participants Achieving American College of Rheumatology 70% (ACR70) Response | Weeks 4, 8, 12, 16, 20 and 24
  ACR70 response: greater than or equal to (>=) 70 percent (%) improvement in painful and tender joint count; >= 70% improvement in swollen joint count; and >= 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP) at each visit.
Change From Baseline in Disease Activity Score Based on 28-Joints Count-High-Sensitivity C-reactive Protein (DAS28-hsCRP) | Weeks 4, 8, 12, 16, 20 and 24
  Disease Activity Score (DAS) based on a 28 joint count hsCRP consisted of composite numerical score of following variables: tender joint count (TJC28), swollen joint count (SJC28), hsCRP (mg/mL), and participant's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP equals to (=) 0.56*square root (sqrt) (TJC28) plus (+) 0.28*sqrt (SJC28) + 0.36*natural log(hsCRP+1) + 0.014*participant's global assessment of disease activity + 0.96. Scores ranged 0-9.4, where lower scores indicated less disease activity. Change = value at observation minus value at baseline.
Change From Baseline in Clinical Disease Activity Index (CDAI) | Weeks 4, 8, 12, 16, 20 and 24
  CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity as assessed by Multi-dimensional Health Assessment Questionnaire (MDHAQ) subscore, and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined. The range for the CDAI is 0 - 76 with a negative change in CDAI score indicating an improvement in disease activity and a positive change in score indicating a worsening of disease activity.
Changes From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Total Score | Weeks 4, 8, 12, 16, 20 and 24
  HAQ-DI score was an evaluation of the functional status for a participant. The 20-question instrument assessed the degree of difficulty a person had in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0, indicated no difficulty, to 3, indicated inability to perform a task in that area. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range: 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Percent Change From Baseline in Participant's Assessment of Pain Based on Visual Analog Scale (VAS) Score | Weeks 4, 8, 12, 16, 20 and 24
  The participants were asked to assess their level of pain by marking a vertical tick on a 100 mm horizontal VAS scale. The scale ranged from 0-100 mm, where 0 indicated no pain and 100 indicated worst possible pain.
Change From Baseline in Patient's Global Assessment of Arthritis | Weeks 4, 8, 12, 16, 20 and 24
  Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm Visual Analog Scale where 0 = very well and 100 = very poorly. Change = score at observation minus score at baseline.
Change From Baseline in Physician's Global Assessment of Arthritis | Weeks 4, 8, 12, 16, 20 and 24
  Physician Global Assessment of Disease Activity was measured on a 0 to 100 mm Visual Analog Scale (VAS), with 0 mm = no disease activity; very good and 100 mm = worst disease activity; very poor. Change = score at observation minus score at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No